CLINICAL TRIAL: NCT03020316
Title: Peer Mentored Approaches For Men And Women With Coronary Artery Disease ("4Steps")
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1507016382
Record Dates: First submitted 2015-10-26; First posted 2017-01-13 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Subjects will be encouraged to follow-up with their primary physicians.
  Subjects will be informed that they will be periodically contacted by telephone and/or email by the research team for future assessments.
- Peer Mentor & Transcendental Meditation (Active Comparator): Subjects will be assigned a peer mentor (a volunteer with CAD). After initial contact, the peer mentor and subject will be encouraged to communicate at whatever frequency or medium they deem most appropriate. This may include speaking by telephone, personal email or meeting in person. Mentors (and subjects if willing) will be asked to keep a log of such contacts, which will be provided to the study staff at interval reassessments.
  In addition to the peer mentor, subjects will be instructed in transcendental meditation (TM) in the standard manner by a trained TM instructor.
  Interventions: Behavioral: Peer Mentor; Behavioral: Transcendental Meditation
- Peer Mentor (Active Comparator): We are no longer recruiting in this arm.
  Subjects will be assigned a peer mentor (a volunteer with CAD). After initial contact, the peer mentor and subject will be encouraged to communicate at whatever frequency or medium they deem most appropriate. This may include speaking by telephone, personal email or meeting in person. Mentors (and subjects if willing) will be asked to keep a log of such contacts, which will be provided to the study staff at interval reassessments.
  Interventions: Behavioral: Peer Mentor

INTERVENTIONS:
Behavioral: Peer Mentor — A volunteer with a similar disease as the subject
  Arms: Peer Mentor; Peer Mentor & Transcendental Meditation
Behavioral: Transcendental Meditation — A meditation technique
  Arms: Peer Mentor & Transcendental Meditation

SUMMARY:
This study will be a pilot prospective randomized study using a peer mentor with or without Transcendental Meditation as compared to usual care for men and women with a new diagnosis of coronary artery disease (CAD). The study is designed to explore between cohort comparisons of perceived stress and a number of additional outcomes. The results of this pilot study will be used in the design of larger future trials.

The target population is adult men and women with a new diagnosis of CAD made on the basis of a myocardial infarction, coronary revascularization procedure, acute coronary syndrome, or imaging test suggestive of CAD.

The overall hypothesis of this proposal is that the addition of a peer mentor and training in Transcendental Meditation to usual care will improve perceived stress and medication adherence for men and women with newly diagnosed CAD as compared with usual care.

DETAILED DESCRIPTION:
The overall hypothesis of this proposal is that the addition of a peer mentor and training in Transcendental Meditation to usual care will improve perceived stress and medication adherence for men and women with newly diagnosed CAD as compared with usual care.

Participants will be "randomized" into one of two study groups:

Arm 1 - Standard Of Care (SOC) Arm 3 - SOC, assignment of a peer mentor, and the opportunity to receive training in transcendental meditation

We are no longer enrolling in Arm 2 of the study (SOC and subjects addition of a peer mentor).

Subjects will be assessed at baseline, 1 month, 6 months, and 12 months with surveys and assessments.

SOC may include routine outpatient physician assessment, preventive medications with appropriate titration, routine blood draws, advice on lifestyle change, referral to cardiac rehabilitation, use of commercially available medical apps.

Investigation - use of peer mentor and use of transcendental meditation.

1. Peer mentor: These are volunteers with CAD, who will undergo training prior to be assigned a mentee. Content of the training will focus on a review of health counseling, basics of CAD pathophysiology and medications, information on situations where the mentor should advise the subject to contact her doctor, and confidentiality. Mentors are intended to provide psychosocial and limited educational support for subjects.
2. Transcendental meditation (TM). TM is a standardized meditation technique done 20 minutes twice each day while sitting with the eyes closed. Although data are heterogeneous, TM has been demonstrated to reduce blood pressure in several small studies.

ELIGIBILITY:
Inclusion Criteria:

For Participants:

* Men and women aged 18-90
* English speaking
* Newly diagnosed with CAD (myocardial infarction [MI], percutaneous coronary intervention [PCI], coronary artery bypass graft [CABG]), acute coronary syndrome, or any imaging test suggestive of CAD).

For Mentors:

(Male mentors will be paired with male participants, and female mentors will be paired with female participants.)

* Men and women aged 18-90
* English speaking
* Established (greater than 1yr prior to study) diagnosis of CAD (myocardial infarction [MI], percutaneous coronary intervention [PCI], coronary artery bypass graft [CABG] acute coronary syndrome, or imaging test suggestive of CAD).

Exclusion Criteria:

For Participants:

* Previously diagnosed CAD (MI, PCI, CABG, acute coronary syndrome or imaging test suggestive of CAD)
* Inability or unwillingness to provide written consent
* Non-English speaking
* Prior formal training and practice of TM

For Mentors:

* Inability or unwillingness to provide written consent
* Non-English speaking

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-04; Primary Completion 2019-10-06 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Perceived Stress | 52 weeks
  Cohen Perceived Stress Scale (PSS-10)
  Each item is rated on a 5-point scale ranging from never (0) to almost always (4). Positively worded items are reverse scored, and the ratings are summed, with higher scores indicating more perceived stress.
  Total scale range: 0-40. Scores around 13 are considered average. Scores of 20 or higher are considered high stress.

SECONDARY OUTCOMES:
Medication Adherence (ARMS-7) | 52 weeks
  Adherence to Refills and Medication Scale (ARMS-7)
  Total scale range: 7-28; subscale range: 1-4. Scores can be treated as a continuous measure or dichotomized as 7 or >7. Lower scores indicate better adherence.
Medication Adherence (VAS) | 52 weeks
  Visual analog scale for medication adherence
  Total scale range: 0-100%. Higher percentage indicates better adherence.
Depressive Symptoms | 52 weeks
  Center for Epidemiologic Studies Depression Scale (CES-D)
  Total scale range: 0-60. Total score of 16 or higher is considered depressed.
Height | 52 weeks
  Height (m)
Weight | 52 weeks
  Weight (kg)
Blood pressure | 52 weeks
  Blood pressure (mmHg)
Heart rate | 52 weeks
  Heart rate (beats/min)
Waist circumference | 52 weeks
  Waist circumference (cm)
Lipid panel results | 52 weeks
  Total cholesterol, LDL, HDL, triglycerides (mg/dL)
Fasting plasma glucose | 52 weeks
  Fasting plasma glucose levels (mg/dL)
Hospital readmission | 52 weeks
  Was the subject readmitted or not
Changes in physical activity | 52 weeks
  Measured by International Physical Activity Questionnaire (IPAQ)
  Survey does not include a range of possible values. Based on verbal description of activity and participation time, populations are divided into 3 proposed levels of physical activity: inactive, minimally active, and HEPA active.
Number and manner of contacts between participants and mentors | 52 weeks
  Verbal description
Participant feedback about mentorship and TM | 52 weeks
  Verbal description
Participant knowledge about CAD | 52 weeks
  Verbal description

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Peña, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- HeartHealth - Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided